CLINICAL TRIAL: NCT01727167
Title: Effects of Low Level Carbon Monoxide Preconditioning on Human Mitochondrial Biogenesis in Aortic Valve Surgery Patients
Brief Title: CO as a Stimulant for Mitochondrial Biogenesis in Human Cardiac Muscle
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Lack of funding and low accrual.
Sponsor: John J Freiberger (Other)
Responsible Party: Sponsor-Investigator, John J Freiberger, Associate Professor of Anesthesiology, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: Pro00031899
Record Dates: First submitted 2012-11-12; First posted 2012-11-15 (Estimated); Results first posted 2016-05-19 (Estimated); Last update posted 2016-05-19 (Estimated); Status verified 2016-05

CONDITIONS: Cardiac Disease; Mitochondrial Biogenesis; Carbon Monoxide
Keywords: cardiac disease; mitochondrial biogenesis; carbon monoxide
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control Group (Placebo Comparator): This group will breath room air for one hour per day over the course of the three days immediately prior to surgery.
  Interventions: Other: Control
- CO group (Experimental): This group will breath 200 ppm of CO for one hour per day over the course of the three days immediately prior to surgery.
  Interventions: Drug: 200ppm CO for one hour

INTERVENTIONS:
Drug: 200ppm CO for one hour — This is the study intervention. The treatment group will breath 200 ppm of CO for one hour over the three days immediately prior to surgery.
  Other Names: CO exposure
  Arms: CO group
Other: Control — This group will breath room air for one hour per day over the course of the three days immediately prior to surgery.
  Arms: Control Group

SUMMARY:
This study will test if inhalation of Carbon Monoxide (CO) will increase the numbers of mitochondria in heart muscle. Mitochondria are the small components of muscle and other cells that convert fuel and oxygen to the easily usable forms of energy (ATP) that power all cell's activities. Adequate numbers of healthy mitochondria are essential to heart cell function. From animal and other studies we have reason to believe that breathing small amounts of CO will signal the body to increase the numbers of mitochondria in heart cells. We propose to test this theory in heart valve surgery patients by examining a small sample of heart tissue (from the right atrial appendage) that is routinely cut out during the preparation of the patient for cardio-pulmonary bypass and that would otherwise be discarded by the surgeon. Muscle samples from two groups of subjects will be compared. One group will breath CO and the other group will breath room air. If CO is effective, we should notice an increase in the numbers of mitochondria in the group that was exposed to CO compared to the group that breathed room air.

DETAILED DESCRIPTION:
PURPOSE AND OBJECTIVE: Endogenously produced carbon monoxide (CO) is known to act as a physiologic signaling molecule to induce mitochondrial biogenesis. This study will test if low-level CO preconditioning induces myocardial biogenesis in humans and if clinical benefit is derived from it. STUDY ACTIVITIES AND POPULATION: The study is an interventional, prospective, randomized, double-blinded trial with a 2-week follow up period. Forty subjects will be recruited from the population of patients scheduled to undergo elective aortic valve replacement. For safety purposes patients with coronary disease will be excluded. Subjects meeting the inclusion criteria will be randomized to receive either air or air containing CO @ 200ppm as a one-hour inhalational treatment per day over the course of the three days immediately prior to their scheduled operation. Biochemical markers for mitochondrial biogenesis (blood and right atrial tissue) and clinical outcome parameters ( BUN/creatinine, and left ventricular function measured by 2D echo) will be measured in all patients pre and post-operatively. Right atrial tissue samples will be collected from tissue that is routinely excised during placement of venous cannulas for cardiopulmonary bypass. RISK/SAFETY & DATA ANALYSIS: Risks will be those of CO inhalation and blood drawing. The 200ppm dose chosen is within OSHA work place exposure limits and has been used safely in human subjects previously. Data will be analyzed by comparing biogenetic marker levels and clinical parameters pre and post intervention and control to CO treatment group.

ELIGIBILITY:
Inclusion Criteria:

1. Able to consent
2. Competent adult
3. Scheduled to undergo aortic or mitral valve surgery only, not combined valve / revascularization procedures.

Exclusion Criteria:

1. Unable to consent
2. Tobacco use
3. Unanticipated medical diagnoses made at the time of surgery which require further procedures lengthening OR time and complexity above that of AVR alone.
4. Concomitant coronary artery disease.
5. Renal dialysis
6. Hemodynamic instability
7. End stage COPD defined as requiring home oxygen
8. By history any significant exposure to second hand smoke including living with a smoker who smokes indoors or working in a high smoking environment for 8 hours a day or more (i.e. factory or bar) will exclude subject from the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2014-02; Primary Completion 2016-01 (Actual); Study Completion 2016-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Duke Hospital, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No
Only one subject was recruited. Funding was not obtained. The study was cancelled with the Duke IRB 3/16.

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group | CO Group
Started | 1 | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Collected demographic and clinical characteristics are not reported to protect patient anonymity.
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group | CO Group | Total
Number analyzed (Participants) | 0 | 0 | 0
Age, Categorical [Count of Participants; unit: Participants]
Sex: Female, Male [Count of Participants; unit: Participants]

OUTCOME MEASURES:

1. Primary Outcome: Biochemical Markers for Mitochondrial Biogenesis (Blood and Right Atrial Tissue)
Description: Right atrial biochemical markers will be measured one time only, intra-operatively. Blood Biochemical markers will be measured before CO exposure and at intervals up to one week post-operatively
Time Frame: 2 weeks
Population: Molecular data was not collected for the single enrolled participant.
Arm/Group | Control Group | CO Group
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Compare Blood to Right Atrial Tissue Biochemical Markers of Mitochondrial Biogenesis
Description: Biochemical markers in both right atrial tissue and blood will be measured and compared to see if the more easily obtained blood markers accurately describe changes expected in the heart.
Time Frame: on week
Population: Molecular data was not collected for the single enrolled participant.
Arm/Group | Control Group | CO Group
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Arm/Group | Control Group | CO Group
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/0
Other Adverse Events (participants affected / at risk) | 0/1 | 0/0

LIMITATIONS AND CAVEATS:
Terminated study due to low accrual.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes